CLINICAL TRIAL: NCT01734993
Title: A Multicenter, Open-Label Long-Term Extension Study of WA22762 to Evaluate Safety and Efficacy of Subcutaneous Tocilizumab in Patients With Moderate to Severe Rheumatoid Arthritis
Brief Title: A Long-Term Extension Study of WA22762 to Evaluate Safety and Efficacy of Subcutaneous Tocilizumab in Participants With Moderate to Severe Rheumatoid Arthritis (RA).
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML28544
Record Dates: First submitted 2012-11-19; First posted 2012-11-28 (Estimated); Results first posted 2016-11-28 (Estimated); Last update posted 2016-11-28 (Estimated); Status verified 2016-10

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tocilizumab

ARMS (1):
- Tocilizumab (Experimental): Moderate to severe rheumatoid arthritis participants from France, who completed the Week 97 visit of the WA22762 LTE study and considered as responders (defined as having improvement in DAS28 of >1.2 points) will continue tocilizumab treatment within this local LTE study for a maximum of 156 weeks, or until SC TCZ becomes commercially available, whichever occurs first.
  Interventions: Drug: Tocilizumab

INTERVENTIONS:
Drug: Tocilizumab — Participants will receive TCZ 162 milligrams (mg) SC injection once a week.
  Other Names: RoActemra; Actemra

SUMMARY:
This multicenter, open-label, single arm, interventional, long-term extension (LTE) study will evaluate the safety and efficacy of tocilizumab (TCZ, RoActemra/Actemra) in French participants with moderate to severe RA who have completed the Week 97 visit of WA22762 LTE study (NCT01194414) (EudraCT Number 2010-018375-22). Participants from France, who completed the Week 97 visit of the WA22762 LTE study and considered as responders (defined as having improvement in disease activity score based on 28-joint count [DAS28] of greater than [>] 1.2 points) will continue TCZ treatment within this local LTE study for a maximum of 156 weeks of subcutaneous (SC) TCZ treatment, or until SC TCZ becomes commercially available, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* Negative pregnancy test at screening and baseline
* Participants who have completed the 97-week WA22762 LTE study on SC or intravenous (IV) TCZ and who experienced, at any time during WA22762, clinically significant improvement in DAS28 (>1.2 points), and based on the investigator's judgment may continue to benefit from TCZ treatment in this study investigating the SC formulation
* No current or recent adverse events or laboratory findings preventing the use of the study drug dose of TCZ 162 mg SC at baseline visit
* Receiving treatment on an outpatient basis
* Females of childbearing potential and males with female partners of childbearing potential must agree to use reliable means of contraception during the study and for at least 3 months following the last dose of study drug
* Oral corticosteroids and non-steroidal anti-inflammatory drugs (NSAIDS) up to the recommended dose are permitted if on stable dose regimen for greater than and equal to (>/=) 4 weeks prior to baseline
* Permitted non-biological disease-modifying anti-rheumatic drugs (DMARDs) are allowed

Exclusion Criteria:

* Participants who have prematurely withdrawn from the WA22762 LTE study for any reason
* Previous treatment with any cell-depleting therapies, including investigational agents or approved therapies
* Treatment with an anti-tumor necrosis factor (TNF) or anti-interleukin (IL) 1 agent, or a T-cell co stimulation modulator since the last administration of study drug in the WA22762 LTE study
* Immunization with a live/attenuated vaccine since the last administration of study drug in the WA22762 LTE study
* Diagnosis, since last WA22762 visit (Week 97), of rheumatic autoimmune disease other than rheumatoid arthritis; secondary Sjörgen's syndrome with RA is permitted
* Diagnosis, since last WA22762 visit (Week 97), of inflammatory joint disease other than RA
* Uncontrolled disease states, such as asthma or inflammatory bowel disease, where flares are commonly treated with oral or parenteral corticosteroids
* Evidence of serious uncontrolled concomitant disease
* Known active current or history of recurrent infection
* Primary or secondary immunodeficiency (history of or currently active)
* Body weight >150 kilograms (kg)
* Pregnant or lactating women
* Inadequate hematologic, renal or liver function
* History of alcohol, drug or chemical abuse within 1 year prior to screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2012-10; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (6):
- France (6):
  - Bordeaux
  - Montpellier
  - Nantes
  - Paris
  - Strasbourg
  - Toulouse

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 12 participants were screened at 6 sites in France, of which 11 participants were enrolled.
Groups:
- Tocilizumab: Moderate to severe rheumatoid arthritis participants from France who completed the Week 97 visit of the WA22762 long term extension (LTE) study (NCT01194414, EudraCT Number 2010-018375-22) and considered as responders (defined as having improvement in DAS28 of greater than [>] 1.2 points) were administered tocilizumab (TCZ) in this long-term extension study, at a dose of 162 milligrams (mg) as subcutaneous (SC) injection once a week, for a maximum of 156 weeks or until SC TCZ was commercially available, whichever occurred first.
Period: Overall Study
Arm/Group | Tocilizumab
Started | 11
Completed | 9
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Lack of Efficacy | 1

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received at least one dose of study medication.
Groups:
- Tocilizumab: Moderate to severe rheumatoid arthritis participants from France who completed the Week 97 visit of the WA22762 LTE study (NCT01194414, EudraCT Number 2010-018375-22) and considered as responders (defined as having improvement in DAS28 of > 1.2 points) were administered TCZ in this long-term extension study, at a dose of 162 mg as SC injection once a week, for a maximum of 156 weeks or until SC TCZ was commercially available, whichever occurred first.
Arm/Group | Tocilizumab
Number analyzed (Participants) | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.91 (11.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 4

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An adverse event (AE) was defined as any untoward medical occurrence in a participant who was administered a study treatment regardless of whether or not the event has a causal relationship with the treatment. An AE, therefore, could be any unfavorable or unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the study treatment, whether or not related to the treatment. A SAE was any untoward medical occurrence that at any dose resulted in death, was life threatening, required hospitalization or prolongation of hospitalization or resulted in disability/incapacity, and congenital anomaly/birth defect. AEs included SAEs as well as non-serious AEs.
Time Frame: Baseline up to approximately 142 weeks
Population: Safety population
Measure: Number; unit: Percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 11
Percentage of participants
  Any AE | 100
  SAE | 18.2

2. Primary Outcome: Percentage of Participants With AEs and SAEs Related to TCZ
Description: An AE was any untoward medical occurrence attributed to study drug in a participant who received study drug. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. AEs included SAEs as well as non-serious AEs. Causality of AEs based on physician's discretion: certain (AE after drug intake, not explained by other drugs, reaction on drug cessation [DC], relapse on re-intake of drug), probable/likely (AE after drug intake, not explained by other drugs, reaction on DC, no information on re-intake), possible (AE after drug intake, explained by other drugs, no information on DC), unlikely (not related to drug intake time, explained by other drugs). AEs with causality of certain, probable/likely, and possible were considered TCZ related.
Time Frame: Baseline up to approximately 142 weeks
Population: Safety population
Measure: Number; unit: Percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 11
Percentage of participants
  Related AE | 72.7
  Related SAE | 9.1

3. Primary Outcome: Percentage of Participants With Adverse Events of Special Interest (AESIs)
Description: Adverse events of special interest (AESI) for this study included: infections (including opportunistic infections), myocardial infarction/acute coronary syndrome, gastrointestinal perforation and related events, malignancies, anaphylaxis / hypersensitivity reactions, demyelinating disorders, stroke, bleeding events and hepatic events.
Time Frame: Baseline up to approximately 142 weeks
Population: Safety population
Measure: Number; unit: Percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 11
Percentage of participants | 18.2

4. Primary Outcome: Percentage of Participants With AESIs Related to TCZ
Description: AESI for this study included: infections (including opportunistic infections), myocardial infarction/acute coronary syndrome, gastrointestinal perforation and related events, malignancies, anaphylaxis / hypersensitivity reactions, demyelinating disorders, stroke, bleeding events and hepatic events. Percentage of participants with AESI related to the drug were presented. Causality of AESIs based on physician's discretion: certain (AE after drug intake, not explained by other drugs, reaction on DC, relapse on re-intake of drug), probable/likely (AE after drug intake, not explained by other drugs, reaction on DC, no information on re-intake), possible (AE after drug intake, explained by other drugs, no information on DC), unlikely (not related to drug intake time, explained by other drugs). AESIs with causality of certain, probable/likely, and possible were considered TCZ related.
Time Frame: Baseline up to approximately 142 weeks
Population: Safety population
Measure: Number; unit: Percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 11
Percentage of participants | 18.2

5. Primary Outcome: Percentage of Participants With AEs Leading to TCZ Discontinuation, Interruption, or Dose Modification
Description: An AE was any untoward medical occurrence attributed to study drug in a participant who received study drug. Percentage of participants with AE causing drug discontinuation, interruption and increase or decrease in dose of drug was presented.
Time Frame: Baseline up to approximately 142 weeks
Population: Safety Population
Measure: Number; unit: Percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 11
Percentage of participants
  AE Leading to Discontinuation | 9.1
  AE Leading to Interruption | 63.6
  AE Leading to Dose Modification | 0.0

6. Primary Outcome: Percentage of Participants With Clinically Significant Physical Examinations and Vital Signs Abnormalities
Description: Criteria for potentially clinically important (PCI) change in vital signs: heart rate value of less than (<) 40 beats per minute and value greater than (>) 150 beats per minute, systolic blood pressure (SBP) of < 80 or >210 millimeter of mercury (mmHg), diastolic blood pressure (DBP) of <40 or >130 mmHg, body temperature <32 or > 40 degrees Celsius, respiratory rate of <10 or > 50 breaths/minute and criteria for PCI change in physical examination: >/=10% increase or decrease of body weight in kilograms (kg).
Time Frame: Baseline up to approximately 142 weeks
Population: Safety population
Measure: Number; unit: Percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 11
Percentage of participants | 0.0

7. Primary Outcome: Percentage of Participants With Clinically Significant Laboratory Abnormalities
Description: Criteria for laboratory tests clinically significant abnormalities included: hemoglobin, hematocrit and red blood cells (RBCs)(< 0.8*lower limit of normal[LLN]); leucocytes (<0.6/greater than [>]1.5*upper limit of normal [ULN]); platelets (<0.5*LLN></0>1.75*ULN); neutrophils, lymphocytes (<0.8*LLN></0>1.2*ULN); eosinophils, basophils, monocytes (>1.2*ULN); total bilirubin, direct bilirubin, indirect bilirubin (>1.5*ULN); aspartate aminotransferase (AST), alanine aminotransferase (ALT), alkaline phosphatase (>3*ULN), total protein, albumin (<0.8*LLN></0>1.2*ULN); creatinine, urea (>1.3*ULN); glucose (<0.6*LLN></0>1.5*ULN); uric acid (>1.2*ULN); sodium, potassium, chloride, calcium, bicarbonate (<0.9*LLN></0>1.1*ULN); urine RBCs, urine white blood cells (WBCs) (> or equal[=]20 high-powered field), urine bacteria >20 high-powered field. Overall percentage of participants with any clinically significant laboratory abnormality was reported.
Time Frame: Baseline up to approximately 142 weeks
Population: Safety population
Measure: Number; unit: Percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 11
Percentage of participants | 9.1

8. Primary Outcome: Percentage of Participants With Anti-TCZ Antibodies
Time Frame: Baseline up to approximately 142 weeks
Population: Safety population
Measure: Number; unit: Percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 11
Percentage of participants | 0.0

9. Secondary Outcome: Change From Baseline in Disease Activity Score 28 - Erythrocyte Sedimentation Rate (DAS28-ESR) Score
Description: The DAS 28 ESR score is a measure of the participant's disease activity calculated using the tender joint count (TJC) [28 joints], swollen joint count (SJC) [28 joints], patient's global assessment (PtGA) of disease activity (visual analog scale [VAS]: 0 millimeter [mm] = no disease activity to 100 mm=maximum disease activity) and the erythrocyte sedimentation rate (ESR in millimeters per hour [mm/hr]). DAS28 was calculated using following formulas: DAS28-ESR = 0.56*square root (sqrt) (TJC28) + 0.28*sqrt (SJC28) + 0.70*natural logarithm (ln) (ESR) + 0.014*PtGA of disease activity. A total possible score of 0 to approximately 10, with higher score indicating more severe disease activity. Completer last visit: Last visit data for participants who completed the study. Last visit: Last visit data for all participants (including those who discontinued prematurely). Early withdrawal: Data at the time of early withdrawal for those participants who discontinued prematurely.
Time Frame: Baseline (Day 0), Weeks 12, 24, 36, 48, 60, 72, 84, 96, 108, 120, completer last visit (up to Week 120), last visit (up to Week 120), early withdrawal (up to Week 120)
Population: Safety population. Here, 'n' represents the number of participants available for assessment at a given time point.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 11
Units on a scale
  Baseline (n=11) | 1.81 (0.87)
  Change at Week 12 (n=8) | 0.16 (1.59)
  Change at Week 24 (n=9) | -0.14 (1.17)
  Change at Week 36 (n=9) | -0.02 (1.30)
  Change at Week 48 (n=10) | -0.32 (0.93)
  Change at Week 60 (n=10) | -0.33 (1.14)
  Change at Week 72 (n=10) | -0.35 (0.92)
  Change at Week 84 (n=9) | 0.28 (1.23)
  Change at Week 96 (n=9) | -0.36 (1.11)
  Change at Week 108 (n=7) | -0.14 (1.55)
  Change at Week 120 (n=2) | -0.75 (0.88)
  Change at Completer last visit (n=9) | -0.16 (1.19)
  Change at Early withdrawal (n=2) | 2.76 (0.87)
  Change at Last visit (n=11) | 0.38 (1.61)

10. Secondary Outcome: Change From Baseline in Simplified Disease Activity Index (SDAI) Score
Description: The SDAI was calculated as (SJC [28 joints] + TJC [28 joints] + VAS ptGA + VAS physician global assessment of disease activity + C-reactive Protein (CRP) level in milligram/deciliter [mg/dL]). VAS assessments: 0 centimeters (cm)=no disease activity to 10 cm=maximum disease activity. SDAI score ranged from 0 to 86, with higher scores indicating increased disease activity. Completer last visit: Last visit data for participants who completed the study. Last visit: Last visit data for all participants (including those who discontinued prematurely). Early withdrawal: Data at the time of early withdrawal for those participants who discontinued prematurely.
Time Frame: as for outcome 9
Population: Safety population. Here, N (number of participants analyzed) represents the number of participants evaluable for this outcome and 'n' represents the number of participants available for assessment at a given time point.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 5
Units on a scale
  Baseline (n=5) | 7.21 (4.15)
  Change at Week 12 (n=5) | 9.17 (12.63)
  Change at Week 24 (n=2) | 8.48 (7.81)
  Change at Week 36 (n=3) | 4.50 (4.61)
  Change at Week 48 (n=2) | -1.02 (0.23)
  Change at Week 60 (n=2) | -1.02 (1.32)
  Change at Week 72 (n=3) | 4.19 (1.66)
  Change at Week 84 (n=3) | 0.83 (3.43)
  Change at Week 96 (n=3) | 0.60 (4.95)
  Change at Week 108 (n=3) | 5.25 (8.15)
  Change at Week 120 (n=0) | NA (NA) — No participant was evaluable for the specified time point.
  Change at Completer last visit (n=2) | 0.69 (5.02)
  Change at Early withdrawal (n=1) | 17.38 (NA) — Standard deviation data is not applicable since only 1 participant was evaluable at indicated time point.
  Change at Last visit (n=3) | 6.25 (10.27)

11. Secondary Outcome: Change From Baseline in TJC
Description: For TJC a total of 28 joints were assessed. The presence of a tender joint was scored as 1 and absence as 0. Total score is calculated by adding the scores, which is ranging from 0 (best possible score or no tender joint) to 28 (worse possible score or all tender joints). Lower scores indicate no tender joint and higher scores indicate worsening tender joints. Completer last visit: Last visit data for participants who completed the study. Last visit: Last visit data for all participants (including those who discontinued prematurely). Early withdrawal: Data at the time of early withdrawal for those participants who discontinued prematurely.
Time Frame: as for outcome 9
Population: Safety population. Here, 'n' represents the number of participants available for assessment at a given time point.
Measure: Mean (Standard Deviation); unit: Tender Joints
Arm/Group | Tocilizumab
Number analyzed (Participants) | 11
Tender Joints
  Baseline (n=11) | 1.27 (1.35)
  Change at Week 12 (n=10) | 0.50 (2.27)
  Change at Week 24 (n=10) | 1.20 (3.01)
  Change at Week 36 (n=10) | 1.00 (1.89)
  Change at Week 48 (n=10) | 0.50 (1.84)
  Change at Week 60 (n=10) | 1.20 (5.31)
  Change at Week 72 (n=10) | 0.60 (3.06)
  Change at Week 84 (n=9) | 0.44 (1.51)
  Change at Week 96 (n=9) | 0.11 (1.27)
  Change at Week 108 (n=7) | 1.57 (5.68)
  Change at Week 120 (n=2) | 0.00 (1.41)
  Change at Completer Last Visit (n=9) | -0.44 (1.24)
  Change at Early Withdrawal n=2) | 6.50 (0.71)
  Change at Last Visit (n=11) | 0.82 (3.03)

12. Secondary Outcome: Change From Baseline in SJC
Description: For SJC, a total of 28 joints were assessed. The presence of a swollen joint was scored as 1 and absence as 0. Total score is calculated by adding the scores, which is ranging from 0 (best possible score or no swollen joint) to 28 (worse possible score or all swollen joints). Lower scores indicate no swollen joint and higher scores indicate worsening swollen joints. Completer last visit: Last visit data for participants who completed the study. Last visit: Last visit data for all participants (including those who discontinued prematurely). Early withdrawal: Data at the time of early withdrawal for those participants who discontinued prematurely.
Time Frame: as for outcome 9
Population: Safety population. Here, 'n' represents the number of participants available for assessment at a given time point.
Measure: Mean (Standard Deviation); unit: Swollen Joints
Arm/Group | Tocilizumab
Number analyzed (Participants) | 11
Swollen Joints
  Baseline (n=11) | 1.00 (1.67)
  Change at Week 12 (n=10) | 0.50 (2.37)
  Change at Week 24 (n=10) | -0.50 (1.84)
  Change at Week 36 (n=10) | -0.60 (2.22)
  Change at Week 48 (n=10) | -0.80 (1.75)
  Change at Week 60 (n=10) | -0.70 (1.49)
  Change at Week 72 (n=10) | -0.30 (2.31)
  Change at Week 84 (n=9) | -0.78 (1.09)
  Change at Week 96 (n=9) | -0.67 (1.41)
  Change at Week 108 (n=7) | 0.14 (2.48)
  Change at Week 120 (n=2) | -0.50 (0.71)
  Change at Completer Last Visit (n=9) | -0.56 (2.24)
  Change at Early Withdrawal (n=2) | 3.5 (2.12)
  Change at Last Visit (n=11) | 0.18 (2.68)

13. Secondary Outcome: Percentage of Participants With Clinical Remission
Description: Clinical remission defined as:DAS28-ESR score < 2.6 and/or SDAI score </= 3.3.DAS28 score is measure of subject's disease activity calculated using TJC [28 joints],SJC [28 joints],PtGA of disease activity [ VAS:0mm= no disease activity to 100 mm=maximum disease activity] and ESR (mm/hr). DAS28 was calculated as DAS28-ESR = 0.56*sqrt (TJC28) + 0.28*sqrt(SJC28) + 0.70* ln ESR + 0.014*PtGA of disease activity. DAS28-ESR score ranged from 0 to approximately 10, higher score indicating more severe disease activity. SDAI was calculated =[SJC (28 joints) + TJC (28 joints) + VAS PtGA + VAS physician global assessment of disease activity+CRP level(mg/dL)]. VAS assessments:0 mm=no disease activity to 100 mm=maximum disease activity. SDAI score ranged from 0 to 86, with higher scores indicating increased disease activity.
Time Frame: Week 48, 108
Population: as for outcome 10
Measure: Number; unit: Percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 10
Percentage of participants
  Week 48 (n=10) | 90
  Week 108 (n=8) | 75

14. Secondary Outcome: Percentage of Participants With Concomitant Corticosteroid Discontinuation
Time Frame: Baseline up to approximately 142 weeks
Population: Safety population. Here, N (number of participants analyzed) represents the participants who received concomitant corticosteroids.
Measure: Number; unit: Percentage of participants
Groups:
- Tocilizumab: Moderate to severe rheumatoid arthritis participants from France who completed the Week 97 visit of the WA22762 LTE study (NCT01194414, EudraCT Number 2010-018375 -22) and considered as responders (defined as having improvement in DAS28 of > 1.2 points) were administered TCZ in this long-term extension study, at a dose of 162 mg as SC injection once a week, for a maximum of 156 weeks or until SC TCZ was commercially available, whichever occurred first.
Arm/Group | Tocilizumab
Number analyzed (Participants) | 6
Percentage of participants | 16.7

15. Secondary Outcome: Percentage of Participants With Concomitant Corticosteroid Dose Reduction
Time Frame: Baseline up to approximately 142 weeks
Population: as for outcome 14
Measure: Number; unit: Percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 6
Percentage of participants | 50

16. Secondary Outcome: Time to Concomitant Corticosteroid Discontinuation
Description: Time to corticosteroid discontinuation = (End date of corticosteroid treatment - date of first drug intake of this extension study) + 1.
Time Frame: Baseline up to approximately 142 weeks
Population: Safety population. Here N (number of participants analyzed) represents the participants who discontinued concomitant corticosteroids
Measure: Median (Full Range); unit: Days
Arm/Group | Tocilizumab
Number analyzed (Participants) | 1
Days | 472.00

17. Secondary Outcome: Time to Concomitant Corticosteroid Dose Reduction
Description: Time to corticosteroid dose reduction (days) = (Date of the first dose reduction of corticosteroid treatment - date of first drug intake of this extension study) + 1.
Time Frame: Baseline up to approximately 142 weeks
Population: Safety population. Here, N (number of participants analyzed) represents the participants who had concomitant corticosteroid dose reduction.
Measure: Median (Full Range); unit: Days
Arm/Group | Tocilizumab
Number analyzed (Participants) | 3
Days | 75 [15.0 to 758.0]

18. Secondary Outcome: Change From Baseline in PtGA of Disease Activity
Description: PtGA of disease activity over the previous 24 hours using a 100 mm VAS where left end of the line 0 mm =no disease activity and right end of the line 100 mm =maximum disease activity. Completer last visit: Last visit data for participants who completed the study. Last visit: Last visit data for all participants (including those who discontinued prematurely). Early withdrawal: Data at the time of early withdrawal for those participants who discontinued prematurely.
Time Frame: as for outcome 9
Population: Safety population. Here, 'n' represents the number of participants available for assessment at a given time point.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Tocilizumab
Number analyzed (Participants) | 11
mm
  Baseline (n=11) | 17.55 (21.06)
  Change at Week 12 (n=11) | 11.82 (36.19)
  Change at Week 24 (n=10) | 4.00 (12.54)
  Change at Week 36 (n=10) | 0.90 (26.82)
  Change at Week 48 (n=9) | -4.89 (14.16)
  Change at Week 60 (n=9) | -0.89 (20.75)
  Change at Week 72 (n=9) | -4.44 (17.54)
  Change at Week 84 (n=9) | 0.22 (16.17)
  Change at Week 96 (n=9) | -3.11 (16.51)
  Change at Week 108 (n=7) | -5.00 (24.21)
  Change at Week 120 (n=2) | -21.50 (23.33)
  Change at Completer last visit (n=8) | -6.38 (14.48)
  Change at Early withdrawal (n=2) | 34.00 (15.56)
  Change at Last visit (n=10) | 1.70 (21.90)

19. Secondary Outcome: Change From Baseline in Patient's Assessment of Pain
Description: Patient's assessment of pain over the previous 24 hours: using a VAS, left end of the line 0 mm=no pain to right end of the line 100 mm=unbearable pain. Completer last visit: Last visit data for participants who completed the study. Last visit: Last visit data for all participants (including those who discontinued prematurely). Early withdrawal: Data at the time of early withdrawal for those participants who discontinued prematurely.
Time Frame: as for outcome 9
Population: Safety Population. Here, 'n' represents the number of participants available for assessment at a given time point.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Tocilizumab
Number analyzed (Participants) | 11
mm
  Baseline (n=11) | 19.18 (20.58)
  Change at Week 12 (n=11) | 10.91 (36.68)
  Change at Week 24 (n=10) | 3.80 (14.99)
  Change at Week 36 (n=10) | -1.90 (20.00)
  Change at Week 48 (n=9) | -6.44 (11.57)
  Change at Week 60 (n=9) | -3.78 (15.63)
  Change at Week 72 (n=9) | -8.11 (16.56)
  Change at Week 84 (n=9) | 0.11 (14.44)
  Change at Week 96 (n=9) | -8.22 (13.22)
  Change at Week 108 (n=7) | -7.86 (18.21)
  Change at Week 120 (n=2) | -20.00 (26.87)
  Change at Completer last visit (n=8) | 1.50 (29.71)
  Change at Early withdrawal (n=2) | 34.50 (16.26)
  Change at Last visit (n=10) | 8.10 (30.16)

20. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire-Disability Index (HAQ-DI) Total Score
Description: The HAQ-DI questionnaire measures functional status (disability) and health-related quality of life. It measures the participant's ability to perform everyday tasks. The index consists of 20 questions regarding the function of the upper and lower extremities. These questions are summarized in 8 categories: dressing and grooming, arising, eating, walking, hygiene, reach, grip, and common activities over past week. Each question is evaluated according to the degree of severity on a 4-point scale. Total score for HAQ-DI was the average of all questions and ranges from 0 = without any difficulty to 3 = unable to do. Completer last visit: Last visit data for participants who completed the study. Last visit: Last visit data for all participants (including those who discontinued prematurely). Early withdrawal: Data at the time of early withdrawal for those participants who discontinued prematurely.
Time Frame: as for outcome 9
Population: Safety population, Here, N (number of participants analyzed) represents the participants who were evaluable for this outcome and 'n' represents the number of participants available for assessment at a given time point.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 7
Units on a scale
  Baseline (n=7) | 0.77 (0.55)
  Change at Week 12 (n=7) | -0.20 (0.52)
  Change at Week 24 (n=7) | 0.18 (0.24)
  Change at Week 36 (n=7) | -0.07 (0.31)
  Change at Week 48 (n=7) | 0.00 (0.54)
  Change at Week 60 (n=7) | -0.13 (0.35)
  Change at Week 72 (n=6) | -0.25 (0.41)
  Change at Week 84 (n=5) | -0.18 (0.62)
  Change at Week 96 (n=5) | 0.08 (0.07)
  Change at Week 108 (n=5) | -0.15 (0.57)
  Change at Week 120 (n=1) | 0.00 (NA) — Standard deviation data is not applicable since only 1 participant was evaluable at indicated time point.
  Change at Completer Last Visit (n=6) | 0.10 (0.43)
  Change at Early Withdrawal (n=1) | 0.00 (NA) — Standard deviation data is not applicable since only 1 participant was evaluable at indicated time point.
  Change at Last Visit (n=7) | 0.09 (0.39)

21. Secondary Outcome: Change From Baseline in Physician's Global Assessment of Disease Activity
Description: The Physician's Global Assessment of disease activity was assessed using a 0 to 100 mm horizontal VAS. The left-hand extreme of the line equals 0 mm, and is described as "no disease activity" (symptom-free and no arthritis symptoms) and the right-hand extreme equals 100 mm, as "maximum disease activity". Completer last visit: Last visit data for participants who completed the study. Last visit: Last visit data for all participants (including those who discontinued prematurely). Early withdrawal: Data at the time of early withdrawal for those participants who discontinued prematurely.
Time Frame: as for outcome 9
Population: Safety population. Here, N (number of participants analyzed) represents the participants who were evaluable for this outcome and 'n' represents the number of participants available for assessment at a given time point.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Tocilizumab
Number analyzed (Participants) | 10
mm
  Baseline (n=10) | 11.00 (10.84)
  Change at Week 12 (n=10) | 17.60 (31.71)
  Change at Week 24 (n=9) | 5.22 (12.37)
  Change at Week 36 (n=9) | 2.22 (17.23)
  Change at Week 48 (n=9) | -4.11 (7.10)
  Change at Week 60 (n=8) | -2.13 (6.06)
  Change at Week 72 (n=8) | -0.75 (7.87)
  Change at Week 84 (n=9) | 1.22 (9.80)
  Change at Week 96 (n=8) | 2.00 (19.25)
  Change at Week 108 (n=7) | 1.00 (6.90)
  Change at Week 120 (n=2) | 2.5 (7.78)
  Change at Completer last visit (n=7) | 6.71 (13.0)
  Change at Early withdrawal (n=2) | 36.5 (10.61)
  Change at Last visit (n=9) | 13.33 (17.70)

22. Secondary Outcome: Change From Baseline in ESR
Description: Blood samples were collected for ESR, which is an acute phase reactant and provides a non-specific measure of inflammation. The test assesses the rate at which red blood cells fall in a test tube. Normal range is 0-30 millimeters per hour (mm/hr). A decrease in the level indicates reduction in inflammation and therefore improvement. Completer last visit: Last visit data for participants who completed the study. Last visit: Last visit data for all participants (including those who discontinued prematurely). Early withdrawal: Data at the time of early withdrawal for those participants who discontinued prematurely.
Time Frame: as for outcome 9
Population: Safety population. Here, 'n' represents the number of participants available for assessment at a given time point.
Measure: Mean (Standard Deviation); unit: mm/hr
Arm/Group | Tocilizumab
Number analyzed (Participants) | 11
mm/hr
  Baseline (n=11) | 5.82 (7.26)
  Change at Week 12 (n=9) | -2.44 (8.34)
  Change at Week 24 (n=9) | -3.11 (8.30)
  Change at Week 36 (n=9) | 1.89 (17.22)
  Change at Week 48 (n=10) | 0.90 (10.21)
  Change at Week 60 (n=10) | -0.10 (12.64)
  Change at Week 72 (n=10) | -2.60 (7.66)
  Change at Week 84 (n=10) | 2.80 (11.82)
  Change at Week 96 (n=9) | -1.22 (9.97)
  Change at Week 108 (n=7) | 3.29 (21.34)
  Change at Week 120 (n=2) | -0.50 (0.71)
  Change at Completer last visit (n=9) | 2.22 (6.55)
  Change at Early withdrawal (n=2) | 14.00 (15.56)
  Change at Last visit (n=11) | 4.36 (9.01)

23. Secondary Outcome: Change From Baseline in CRP
Description: Blood samples were collected for CRP, which is an acute phase reactant and a measure of inflammation. Completer last visit: Last visit data for participants who completed the study. Last visit: Last visit data for all participants (including those who discontinued prematurely). Early withdrawal: Data at the time of early withdrawal for those participants who discontinued prematurely.
Time Frame: as for outcome 9
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: milligrams per liter (mg/L)
Arm/Group | Tocilizumab
Number analyzed (Participants) | 5
milligrams per liter (mg/L)
  Baseline (n=5) | 0.49 (0.47)
  Change at Week 12 (n=5) | 1.07 (2.17)
  Change at Week 24 (n=2) | -0.25 (0.35)
  Change at Week 36 (n=3) | -0.02 (0.52)
  Change at Week 48 (n=3) | -0.05 (0.65)
  Change at Week 60 (n=3) | -0.09 (0.66)
  Change at Week 72 (n=3) | -0.05 (0.61)
  Change at Week 84 (n=3) | -0.05 (0.51)
  Change at Week 96 (n=3) | -0.02 (0.62)
  Change at Week 108 (n=3) | 1.55 (2.13)
  Change at Week 120 (n=0) | NA (NA) — No participant was evaluable for the specified time point.
  Change at Completer last visit (n=3) | 0.01 (0.54)
  change at Early withdrawal (n=1) | 4.79 (NA) — Standard deviation data is not applicable since only 1 participant was evaluable at indicated time point.
  Change at Last visit (n=4) | 1.21 (2.43)

ADVERSE EVENTS:
Time Frame: Baseline up to approximately 142 weeks
Arm/Group | Tocilizumab
Serious Adverse Events (participants affected / at risk) | 2/11
Other Adverse Events (participants affected / at risk) | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tocilizumab (N=11)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1
Inflammatory pseudotumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Extremity necrosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tocilizumab (N=11)
Bronchitis (Infections and infestations) | 5
Urinary tract infection (Infections and infestations) | 3
Nasopharyngitis (Infections and infestations) | 2
Rhinitis (Infections and infestations) | 2
Sinusitis (Infections and infestations) | 2
Gastroenteritis (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Oral herpes (Infections and infestations) | 1
Tooth infection (Infections and infestations) | 1
Vulvovaginal mycotic infection (Infections and infestations) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 4
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Rheumatoid nodule (Musculoskeletal and connective tissue disorders) | 1
Sjogren's syndrome (Musculoskeletal and connective tissue disorders) | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Dental caries (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Radicular cyst (Gastrointestinal disorders) | 1
Dacryostenosis acquired (Eye disorders) | 1
Eye pruritus (Eye disorders) | 1
Ocular hyperaemia (Eye disorders) | 1
General physical health deterioration (General disorders) | 1
Injection site erythema (General disorders) | 1
Pain (General disorders) | 1
Pyrexia (General disorders) | 1
Ligament sprain (Injury, poisoning and procedural complications) | 1
Limb injury (Injury, poisoning and procedural complications) | 1
Lip injury (Injury, poisoning and procedural complications) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Scan abdomen abnormal (Investigations) | 1
Lipid metabolism disorder (Metabolism and nutrition disorders) | 1
Benign neoplasm of spinal cord (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pyelocaliectasis (Renal and urinary disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 1
Tooth extraction (Surgical and medical procedures) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.